CLINICAL TRIAL: NCT04638166
Title: Mineral Water for Prevention of Renal Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MINERVA
Record Dates: First submitted 2020-10-25; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Calcium Oxalate Urolithiasis
Keywords: Mineral water; Disease prevention; 24h urine analysis
MeSH Terms: conditions — Nephrolithiasis, Calcium Oxalate | interventions — Mineral Waters

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mineral water group (Experimental): The mineral water group were instructed to consume 1.25L of a commercially supplied bicarbonate rich mineral water per day at meal times, supplemented by other fluid intake up to 2.5 - 3L/day.
  Interventions: Other: Mineral water
- Plain water group (Active Comparator): The plain water group consumed only plain water up to 2.5 - 3L/day.
  Interventions: Other: Plain water

INTERVENTIONS:
Other: Mineral water — Drinking mineral water for 12 weeks
  Arms: Mineral water group
Other: Plain water — Drinking plain water for 12 weeks
  Arms: Plain water group

SUMMARY:
The investigators would like to assess if the intake of high bicarbonate mineral water would not only increase total fluid intake but will also be able to give patients the additional benefit of correcting the urinary abnormalities which may predispose them to stone formation.

DETAILED DESCRIPTION:
The life time risk of developing nephrolithiasis is about 10-15% in the western world, but can be as high as 20-25% in the middle east. Evidence suggests that the incidence and prevalence of kidney stones is increasing globally which represent a significant economic burden. Besides the lack of hydration, the most common metabolic abnormalities associated with calcium stones are hypercalciuria, hypocitraturia and hyperoxaluria. In addition, low urinary pH from consumption of non-dairy animal protein has been associated with reduced urinary citrate and increased uric acid stones which form a nidus for subsequent calcium oxalate precipitates.

Dietary modification is the first line approach in the treatment of idiopathic calcium oxalate (CaOx) nephrolithiasis. General advice includes adequate hydration, avoiding oxalate-rich foods, and consumption of an adequate amount of calcium. Adequate hydration is an easy and effective way of preventing stones. Siener et al found in healthy men, consumption of mineral water rich in magnesium and bicarbonate resulted in favourable changes in urinary pH, magnesium and citrate excretion (inhibitors of CaOx stone formation). Our pilot study in 10 young and healthy surgical residents also revealed similar results after drinking bicarbonate rich mineral water for 1 week.

In this study, the investigators compared the effect of drinking bicarbonate rich mineral water with plain water on urine biochemistry in a prospective randomized study in patients with known CaOx stones. The investigators hypothesize that the intake of bicarbonate rich mineral water, particularly at meal times, reduces stone risk via reduction in urinary oxalate through increased intestinal oxalate binding with dietary calcium. Other potential benefits of mineral water include increased urinary stone inhibitors like magnesium, citrate and alkalinisation of urine.

ELIGIBILITY:
Inclusion Criteria:

* patients with proven Calcium Oxalate (CaOx) stone (CaOx >50% by infrared spectroscopy) from Jan 2018 to Aug 2019 in Singapore General Hospital
* all stone formers had suffered spontaneous passage or surgical removal of a urinary calculus during the study period.

Exclusion Criteria:

* presence of urinary tract infection
* severe cardiovascular insufficiency
* previously diagnosed causal metabolic disease such as hyperparathyroidism, renal tubular acidosis, primary hyperoxaluria, Wilson's disease, Cushing disease, osteoporosis and malignant diseases.
* pregnant women
* chronic intestinal diseases
* history of previous bowel resection
* participation in competitive sports

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
changes of Tiselius Index | 1, 4, 8 and 12 weeks
  compare Tiselius Index (24h urine analysis) at week 1, 4, 8 and 12 to baseline (week 0)
changes of urinary oxalate level (mmol/24h) | 1, 4, 8 and 12 weeks
  compare urinary oxalate level (24h urine analysis) at week 1, 4, 8 and 12 to baseline (week 0)

SECONDARY OUTCOMES:
changes of other stone inhibitor/promoter (mmol/24h) | 1, 4, 8 and 12 weeks
  compare Magnesium, Citrate, Sodium, Calcium, Uric Acid (24h urine analysis) at week 1, 4, 8 and 12 to baseline (week 0)
changes of urinary volume (ml/24h) | 1, 4, 8 and 12 weeks
  compare urinary volume (24h urine analysis) at week 1, 4, 8 and 12 to baseline (week 0)
changes of urinary pH | 1, 4, 8 and 12 weeks
  compare urinary pH (24h urine analysis) at week 1, 4, 8 and 12 to baseline (week 0)
changes of serum electrolytes (mmol/L) | 12 weeks
  compare serum sodium, potassium, calcium, phosphate, bicarbonate and uric acid at baseline (week 0) and the end of the study (week 12)

CONTACTS AND LOCATIONS:
Overall Officials: Tsung Wen Chong, MBBS, PhD, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No